CLINICAL TRIAL: NCT05940935
Title: The Relationship of Developing Metabolic Acidosis With Antiepleptic Drugs in Craniotomy Operations; Does Topiramat or Zonisamide Cause Metabolic Acidosis?
Brief Title: The Relationship of Developing Metabolic Acidosis With Antiepleptic Drugs in Craniotomy Operations
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation, Principal Investigator, Resident Doctor, Trakya University
Other Study IDs: TÜTF-GOBAEK 2023/210
Record Dates: First submitted 2023-06-21; First posted 2023-07-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Acidosis; Antiepileptic Drugs; Craniotomy; Anesthesia Management
Keywords: Antiepileptic Drugs; Metabolic Acidosis; Anesthesia Management; Craniotomy
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Patients who have used Zonisamide or Topiramate
  Interventions: Procedure: Arterial Blood Gas Base Deficit
- Group 2: Patients who have used Lacosamide
  Interventions: Procedure: Arterial Blood Gas Base Deficit
- Group 3: Patients who have used Carbamazepine
  Interventions: Procedure: Arterial Blood Gas Base Deficit
- Group 4: Patients who have used levetiracetam
  Interventions: Procedure: Arterial Blood Gas Base Deficit

INTERVENTIONS:
Procedure: Arterial Blood Gas Base Deficit — The base deficit values in the preoperative, intraoperative and postoperative blood gases taken from the patients and the presence and severity of metabolic acidosis were evaluated. Metabolic acidosis severity was defined by base deficit levels: mild from -3 to -5, moderate from -5 to -10, and severe metabolic acidosis below -10.

SUMMARY:
The relationship of developing metabolic acidosis with antiepleptic drugs in craniotomy operations

DETAILED DESCRIPTION:
Metabolic acidosis is a life-threatening complication in the perioperative, intraoperative and postoperative period. It can cause decreased cardiac output, electrolyte imbalance, surgical bleeding and neurological complications, even coma and death in surgical patients.

Topiramate and zonisamide are sulfonamide derivative compounds used in the treatment of epilepsy. It has been shown in studies that both drugs have a strong inhibition of carbonic anhydrase enzyme. Recent case reports suggest that both drugs may cause metabolic acidosis by lowering serum bicarbonate levels in some patients.

Aim in this study is to determine the relationship between preoperative, intraoperative and postoperative metabolic acidosis and to emphasize the importance of anesthesia management in patients who have undergone craniotomy and use antiepileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing intracranial surgery with craniotomy and using antiepileptic drugs
* ASA I-III
* Patients undergoing elective surgery

Exclusion Criteria:

* Patients with a surgical procedure time of more than 5 hours
* Patients who received more than 2 units of blood transfusion during the operation
* Patients taking other drugs that can cause metabolic acidosis
* Patients with diabetes mellitus, diabetes insipidus, hepatic or renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent craniotomy and intracranial surgery at Trakya University Medical Faculty Hospital and used antiepileptic drugs were included in the study as a retrospective file review. The files of 35 patients who met the study criteria were reviewed retrospectively.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Preoperative Metabolic Acidosis | Baseline
  The base deficit values in the preoperative, intraoperative and postoperative blood gases taken from the patients and the presence and severity of metabolic acidosis were evaluated. Metabolic acidosis severity was defined by base deficit levels: mild from -3 to -5, moderate from -5 to -10, and severe metabolic acidosis below -10.
Intraoperative Metabolic Acidosis | during the operation
  The base deficit values in the preoperative, intraoperative and postoperative blood gases taken from the patients and the presence and severity of metabolic acidosis were evaluated. Metabolic acidosis severity was defined by base deficit levels: mild from -3 to -5, moderate from -5 to -10, and severe metabolic acidosis below -10.
Postoperative Metabolic Acidosis | Day 1
  The base deficit values in the preoperative, intraoperative and postoperative blood gases taken from the patients and the presence and severity of metabolic acidosis were evaluated. Metabolic acidosis severity was defined by base deficit levels: mild from -3 to -5, moderate from -5 to -10, and severe metabolic acidosis below -10.

CONTACTS AND LOCATIONS:
Overall Officials: SEVTAP HEKİMOĞLU ŞAHİN, Professor, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No